CLINICAL TRIAL: NCT02632422
Title: Intermittent Hypoxia-Induced Recovery of Overground Walking in Persons With Subacute SCI
Brief Title: AIH-induced Walking Recovery After Subacute SCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Randy Trumbower, PT, PhD, Assistant Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017P001941
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injury
Keywords: walk; rehabilitation; strength; movement; spinal cord trauma; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Walking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Non-ambulatory - dAIH (Experimental): Non-ambulatory subjects will be randomly assigned to receive 10 sessions of daily acute intermittent hypoxia (dAIH) 10 treatment visits at a frequency of 5 days each week for 2 weeks.
  Interventions: Other: Daily acute intermittent hypoxia (dAIH)
- Non-ambulatory - dSHAM (Sham Comparator): Non-ambulatory subjects will be randomly assigned to receive 10 sessions of daily room air (dSHAM) 10 treatment visits at a frequency of 5 days each week for 2 weeks.
  Interventions: Other: dSHAM
- Ambulatory - dAIH+Walk (Experimental): Ambulatory subjects will be randomly assigned to receive 10 sessions of daily acute intermittent hypoxia (dAIH) coupled with 60 minutes of walking practice at a frequency of 5 days each week for 2 weeks.
  Interventions: Other: Daily acute intermittent hypoxia (dAIH); Other: Walking
- Ambulatory - dSHAM+Walk (Sham Comparator): Ambulatory subjects will be randomly assigned to receive 10 sessions of daily room air (dSHAM) coupled with 60 minutes of walking practice at a frequency of 5 days each week for 2 weeks.
  Interventions: Other: dSHAM; Other: Walking
- Ambulatory-Walk (Other): Ambulatory subjects will be randomly assigned to 10 sessions of walking practice only for 5 consecutive sessions/week x 2 weeks.
  Interventions: Other: Walking

INTERVENTIONS:
Other: Daily acute intermittent hypoxia (dAIH) — Each participant will be exposed to 10 sessions of daily acute intermittent hypoxia (dAIH) via air generators. The generator will fill reservoir bags attached to a non-rebreathing facemask. Each session will consist of 15 episodes which include intervals of 1.5 minute hypoxia (FIO2=0.10±0.02, i.e. 10% O2) and 1 minute normoxia (FIO2=0.21±0.02). Participants will receive 5 consecutive days of daily acute intermittent hypoxia (dAIH).
  Arms: Ambulatory - dAIH+Walk; Non-ambulatory - dAIH
Other: dSHAM — Each participant will be exposed to 10 sessions of daily room air (dSHAM) via air generators. The generator will fill reservoir bags attached to a non-rebreathing facemask. Each session will consist of 15 episodes of 1.5 minute normoxia (FIO2=0.21±0.02). Participants will receive 5 consecutive days of daily room air (dSHAM).
  Arms: Ambulatory - dSHAM+Walk; Non-ambulatory - dSHAM
Other: Walking — Participants will participate in 10 days of walking practice sessions. Walking practice sessions will immediately follow (within 60 minutes) the breathing intervention during training visits and will last for 60 minutes.
  Walking practice will incorporate 5 walking-related tasks:
  1. walking balance (e.g., walking with turns)
  2. skilled walking tasks (e.g., negotiating obstacles)
  3. walking with secondary task (e.g., walking and talking)
  4. endurance
  5. speed
  Arms: Ambulatory - dAIH+Walk; Ambulatory - dSHAM+Walk; Ambulatory-Walk

SUMMARY:
The purpose of this study is to determine how mild breathing bouts of low oxygen may restore walking and leg strength in persons who have sustained a spinal cord injury.

DETAILED DESCRIPTION:
The goal of the study is to determine whether repeatedly breathing mild bouts of low oxygen for brief periods (termed acute intermittent hypoxia (AIH)) improves recovery of walking and strength after spinal cord injury. This idea stems from animal studies on respiration, in which investigators showed that mild AIH improves breathing in rats with spinal injuries. These studies showed that AIH induces plasticity, strengthening neural connections by increasing the production of key proteins and improving the sensitivity of spinal cord circuitry. The ultimate goal of this research is to assess the potential of mild AIH as a therapeutic approach not only in persons with chronic spinal cord injury but also in persons with subacute injury. By applying AIH during early stages of recovery, the investigators hope to expand the potential benefits of AIH to a broader range of persons with spinal injury, thereby improving functional independence and quality of life for servicemen and civilians.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old
* medically stable with medical clearance from physician to participate
* spinal cord injury (SCI) at or below C3 (phrenic sparing) and above L5 with at least motor function preserved below the neurologic level
* non-progressive etiology of spinal injury
* American Spinal Injury Association Impairment Scale (AIS) grade A-D
* 2-12 months post-injury (subacute)

Exclusion Criteria:

* severe concurrent illness or pain, including unhealed decubiti, severe neuropathic or chronic pain syndrome, infection (e.g. bladder), hypertension, cardiovascular disease, pulmonary disease, severe osteoporosis (history of fractures), active heterotopic ossification in the lower extremities, or history of peripheral nerve injury in the legs
* score less than 24 on Mini-Mental Exam
* severe autonomic dysreflexia
* history of cardiovascular/pulmonary complications
* pregnancy
* severe obstructive sleep apnea (OSA), characterized by uncontrolled hypoxia and sleep fractionation

Specific inclusion/exclusion criteria for recruiting non-ambulatory subjects:

Participation in this group requires all of the above inclusion/exclusion criteria, as well as being unable to complete any of the below measures:

* timed up-and-go (TUG) test
* 10-meter walk test (10MWT)
* 6-minute walk test (6MWT)

Specific inclusion/exclusion criteria for recruiting ambulatory subjects:

Participation in this group requires all of the above criteria, as well as successful completion of at least one below measure:

* timed up-and-go (TUG) test
* 10-meter walk test (10MWT)
* 6-minute walk test (6MWT)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in walking recovery, assessed by timed up-and-go (TUG) test | Baseline, Post-session 10 (up to two weeks)
  The TUG test is used to assess the dynamic balance of an individual. It measures the amount of time (recorded in seconds) it takes for the individual to rise from a standard arm chair, walk a distance of 3 meters and return to the initial position resting against the back of the chair. Participants will perform up to three trials of the TUG test. Average speed across TUG trials will be used for analysis. Change is the difference between the end of session 10 and baseline.
Change in walking recovery, assessed by 6 minute walk test (6MWT) | Baseline, Post-session 10 (up to two weeks)
  Participants perform the 6MWT at their fastest, most comfortable walking speed sustainable for 6 minutes. Distances will be recorded at 2 and 6 minutes. The test will be based upon the participant's ability to finish each assessment without human assistance. Change is the difference between the end of session 10 and baseline.
Change in walking recovery, assessed by 10 meter walk test (10MWT) | Baseline, Post-session 10 (up to two weeks)
  Participants walk ten meters without assistance at their fastest, but safest speed with a minimum of 1-minute of rest between two trials. Average speed across the up to three 10MWT trials will be used for analysis. Change is the difference between the end of session 10 and baseline.

SECONDARY OUTCOMES:
Change in pain severity | Baseline, Post-session 10 (up to two weeks)
  Participants will report their pain level using the Wong-Baker FACES scale. The scale is from 0 to 5; 0 being no pain and 5 being extreme pain. Change is the difference between the end of session 10 and baseline.
Change in spasticity | Baseline, Post-session 10 (up to two weeks)
  Spasticity will be assessed using the Spinal Cord Assessment Tool for Spastic Reflexes (SCATS). The study team will quantify the total lower extremity spasticity score using the cumulative sum of 3 SCATS subscales: clonus (0=no spasticity; 3=severe), flexor (0=no spasticity; 3=severe), and extensor (0=no spasticity; 3=severe). Change is the difference between the end of session 10 and baseline.
Systemic hypertension incidence rate | Post-session 10 (up to two weeks)
  Participants will have their systolic and diastolic blood pressure measured. A systemic hypertensive event is quantified as a systolic pressure exceeding 140mmHg and/or diastolic pressure exceeding 90mmHg. A hypertension incident rate is the number of hypertensive events divided by the total person-time. Person-time is in units of person-measures (the sum of the total number of BP measurements) taken for each person. Person-measures accounts for the total number of chances for detecting a hypertensive event and accounts for measurements not made due to drop-out or a disqualifying adverse event
Autonomic dysreflexia incidence rate | Post-session 10 (up to two weeks)
  The occurrence of autonomic dysreflexia will be assessed. An autonomic dysreflexia event will constitute a participant having a systolic blood pressure (SBP) increase from baseline of 20mmHg or SBP greater than 150mmHg with complaints of headache, diaphoresis, and/or blurred vision and will be diagnosed by the study team clinicians.

CONTACTS AND LOCATIONS:
Overall Officials: Randy Trumbower, PT, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (2):
- United States (2):
  - Shepherd Center, Atlanta, Georgia
  - Spaulding Rehabilitation Hospital, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Trumbower RD, Hayes HB, Mitchell GS, Wolf SL, Stahl VA. Effects of acute intermittent hypoxia on hand use after spinal cord trauma: A preliminary study. Neurology. 2017 Oct 31;89(18):1904-1907. doi: 10.1212/WNL.0000000000004596. Epub 2017 Sep 29. PMID 28972191
- [Background] Hayes HB, Jayaraman A, Herrmann M, Mitchell GS, Rymer WZ, Trumbower RD. Daily intermittent hypoxia enhances walking after chronic spinal cord injury: a randomized trial. Neurology. 2014 Jan 14;82(2):104-13. doi: 10.1212/01.WNL.0000437416.34298.43. Epub 2013 Nov 27. PMID 24285617
- [Background] Trumbower RD, Jayaraman A, Mitchell GS, Rymer WZ. Exposure to acute intermittent hypoxia augments somatic motor function in humans with incomplete spinal cord injury. Neurorehabil Neural Repair. 2012 Feb;26(2):163-72. doi: 10.1177/1545968311412055. Epub 2011 Aug 5. PMID 21821826
- [Background] Hayes HB, Chvatal SA, French MA, Ting LH, Trumbower RD. Neuromuscular constraints on muscle coordination during overground walking in persons with chronic incomplete spinal cord injury. Clin Neurophysiol. 2014 Oct;125(10):2024-35. doi: 10.1016/j.clinph.2014.02.001. Epub 2014 Feb 14. PMID 24618214
- [Background] Peters DM, Thibaudier Y, Deffeyes JE, Baer GT, Hayes HB, Trumbower RD. Constraints on Stance-Phase Force Production during Overground Walking in Persons with Chronic Incomplete Spinal Cord Injury. J Neurotrauma. 2018 Feb 1;35(3):467-477. doi: 10.1089/neu.2017.5146. Epub 2017 Oct 27. PMID 28762876
- [Background] Sohn WJ, Tan AQ, Hayes HB, Pochiraju S, Deffeyes J, Trumbower RD. Variability of Leg Kinematics during Overground Walking in Persons with Chronic Incomplete Spinal Cord Injury. J Neurotrauma. 2018 Nov 1;35(21):2519-2529. doi: 10.1089/neu.2017.5538. Epub 2018 Jun 5. PMID 29648987
- [Background] Naidu A, Peters DM, Tan AQ, Barth S, Crane A, Link A, Balakrishnan S, Hayes HB, Slocum C, Zafonte RD, Trumbower RD. Daily acute intermittent hypoxia to improve walking function in persons with subacute spinal cord injury: a randomized clinical trial study protocol. BMC Neurol. 2020 Jul 8;20(1):273. doi: 10.1186/s12883-020-01851-9. PMID 32641012
- [Result] Tan AQ, Papadopoulos JM, Corsten AN, Trumbower RD. An automated pressure-swing absorption system to administer low oxygen therapy for persons with spinal cord injury. Exp Neurol. 2020 Nov;333:113408. doi: 10.1016/j.expneurol.2020.113408. Epub 2020 Jul 17. PMID 32682613
- See also: INSPIRE Lab - mission is to inspire persons with paralysis to move again — http://inspire-lab.org